CLINICAL TRIAL: NCT01741506
Title: Coagulation Profile in Patients Undergoing Video Assisted Thorascopic Surgery (VATS) for Lung Cancer - A Randomized, Controlled Trial
Brief Title: Coagulation Profile in Patients Undergoing Video Assisted Thorascopic Surgery (VATS) for Lung Cancer
Acronym: COPPVATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Decker Christensen (Other)
Responsible Party: Sponsor-Investigator, Thomas Decker Christensen, Senior staff surgeon, MD, DMSc, PhD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COPPVATS vs 1.1; 2012-002409-23 (EudraCT Number)
Record Dates: First submitted 2012-11-25; First posted 2012-12-05 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-04

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Surgery; Thromboembolism; Bleeding
MeSH Terms: conditions — Lung Neoplasms; Thromboembolism; Hemorrhage | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dalteparin (Fragmin®) (Experimental): Dalteparin (Fragmin®) 5000 IU (International Unit) once daily
  Interventions: Drug: Dalteparin (Fragmin®)
- No treatment (No Intervention): No treatment
- Open surgery arm (Other): Dalteparin (Fragmin®) 5000 IU once daily
  Interventions: Drug: Dalteparin (Fragmin®)

INTERVENTIONS:
Drug: Dalteparin (Fragmin®)
  Arms: Dalteparin (Fragmin®); Open surgery arm

SUMMARY:
The purpose of the study is:

To estimate patients with lung cancers who will undergo surgery total haemostatic / thrombotic capacity pre, per-and postoperatively.

To investigate whether prophylactic treatment with Low Molecular Weight Heparin (LMWH) affects the patient's potential hypercoagulability.

To investigate whether there are differences in patients who will undergo Video Assisted Thorascopic Surgery (VATS) or open surgery in regards of impact of the coagulation system.

DETAILED DESCRIPTION:
Lung cancer is a serious and very frequent disease. For those 25% of the patients who will undergo surgery, there are two different methods of operation: either open surgery (thoracotomy) or Video Assisted Thorascopic Surgery (VATS). The latter method is increasing in use.

Patients are often prescribed heparin pre- postoperatively, but it is unclear whether this prophylactic treatment is necessary, and it has never been thoroughly investigated.

When patients receive heparin there is an increased risk of bleeding.

Furthermore, it is unclear what changes occurs in the coagulation system pre, per- and postoperatively in patients undergoing surgery for lung-cancer, and hereby it is unclear whether these patients should have some sort of medical prophylactic treatment.

By using new analysis methods in terms of Thromboelastometry, Thrombin generation and thrombocyte function analysis, hereby the total coagulation profile can be characterized and hereby estimate the risk of thrombosis and bleeding. Thereby better be able to give the right treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergo surgery for lung cancer with an expected lobectomy or bilobectomy
* The surgery shall be VATS (for patients in the group randomized to other low molecular weight heparin and no prophylactic)
* Willing to be randomized (VATS-patients)
* Over 18 years old.
* Able to give assigned informed consent
* Women should be prescribed secure anticonception.

Exclusion Criteria:

* Thromboembolic events within the last three months (both venous and arterial)
* Pregnant
* Lactating
* Treatment with anticoagulation therapy in terms of vitamin K antagonist or direct or indirect thrombin inhibitors (dabigatran, apixaban or rivaroxaban)
* Treatment with thrombocyte function inhibitors in terms of Clopidogrel, ASA (acetylsalicylic acid), prasugrel and ticagrelor, and no pause of minimum 5 days (7 days with regards of prasugrel) before surgery
* Allergy for LMWH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Thromboelastometry (ROTEM®) | 30 days
  Analysis of in-tem, ex-tem, fib-tem og hep-tem and estimation of: Clotting time (CT (sec)), propagation (MaxVel (mm*100/sec) t,MaxVel, s) og termination (maximum clot firmness (MCF)(mm*100/sec)

SECONDARY OUTCOMES:
Thrombin generation | 30 days
  1) recalcificering, 2) activation with tissue factor 1:17,000 and estimation of Lag time [min], ETP (endogenous thrombin potential) [nM (nanomole) thrombin*minute], peak levels of thrombin generation [nM thrombin] and time to peak thrombin (ttpeak) [min].

OTHER OUTCOMES:
Standard coagulation analysis | 30 days
  APTT (activated partial thromboplastin time), INR (International Normalized Ratio), fibrinogen, fibrin d-dimer, thrombin time, thrombocytes and Factor VIII: clot.
Thrombocyte function analysis | 30 days
  analysis on Multiplate®, where the thrombocyte aggregation are expressed as Aggregation unit (AU), area under curve (A*min).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Christensen, MD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Christensen TD, Vad H, Pedersen S, Licht PB, Nybo M, Hornbech K, Zois NE, Hvas AM. Video-assisted Thoracoscopic surgery (VATS) lobectomy for lung cancer does not induce a procoagulant state. Thromb J. 2017 Dec 20;15:29. doi: 10.1186/s12959-017-0152-2. eCollection 2017. PMID 29270080